CLINICAL TRIAL: NCT03873142
Title: The Effectiveness of a Mindful Parenting Intervention for Parents of Children With Psoriasis and Parents of Children With Eczema: A Single Group Case Series
Brief Title: The Effectiveness of a Mindful Parenting Intervention for Parents of Children With Psoriasis and Parents of Children With Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: The Psoriasis and Psoriatic Arthritis Alliance (Unknown)
Responsible Party: Principal Investigator, Andrew Thompson, Principal Investigator, University of Sheffield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 249150
Record Dates: First submitted 2019-03-04; First posted 2019-03-13 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis; Eczema; Stress
MeSH Terms: conditions — Psoriasis; Eczema

STUDY DESIGN:
Intervention Model Description: A single-group case-series design will be adopted, whereby one group of participants will complete daily and weekly measures over the course of 1) a 2-week baseline period; 2) an 8-week intervention period; 3) an 8-week follow up period. Variables collected during the intervention and follow-up period will be compared with those from the baseline period.
Masking Description: No party will be masked in this study. There is only one arm and participants will act as their own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful parenting intervention (Experimental): There is only one arm in this study. A range of variables will first be measured (daily and weekly) over a baseline period in a group of participants. Following this baseline period, participants will be take part in a mindful parenting intervention whilst the same variables are measured. Following the intervention, there will be an 8-week follow-up period, and mindful parenting groups will not run during this time.
  Interventions: Behavioral: Mindful Parenting

INTERVENTIONS:
Behavioral: Mindful Parenting — The mindful parenting intervention is an adaption for parents of the Mindfulness-Based Cognitive Therapy (MBCT) for depression (Kabat-Zinn, 1990), and the Mindful-Based Stress Reduction program (MBSR; Kabat-Zinn, 1990). The mindful parenting intervention will follow the manual developed by Bögels and Restifo (2014). The intervention consists of 9x3hour sessions. Eight of these sessions are run on consecutive weeks and the final session is run eight weeks after the eighth session. These groups involve group discussions around parenting, meditation exercises, and yoga, amongst other things.

SUMMARY:
This study investigates the impact of a mindful parenting intervention on parents of children with psoriasis or eczema. More specifically, this study will investigate the impact of the group on both the child and the parents mental health and quality of life.

DETAILED DESCRIPTION:
Psoriasis and eczema are chronic inflammatory skin conditions that affect up to 2% and 20% of children respectively (Mahe, 2016; Plötz, Wiesender, Todorva & Ring, 2014). These skin conditions are associated with poorer mental health in the children themselves and in their parents (Megna et al., 2015; Hammer-Helmich et al., 2016). Little research has investigated ways of reducing parental stress in parents of children with chronic health conditions, such as psoriasis and eczema.

"Mindful Parenting" interventions offer one potential way of improving mental health and quality of life in parents and their children. Mindful parenting refers to a parenting style which involves paying close, non-judgemental attention to the child (Duncan et al., 2009). However, no research has investigated the impact of mindful parenting interventions on children with skin conditions and their parents.

The main aim of the current study is to investigate whether a mindful parenting intervention can improve mental health and quality of life in children with psoriasis/eczema and their parents. A single-group case-series design will be adopted, whereby participants will act as their own control; data collected from participants during and after they have received the intervention will be compared to data collected before they have received the intervention. Interviews will also be conducted after the intervention, to explore participants experience of the group.

The investigators predict that the intervention will improve mental health and quality of life in children with psoriasis/eczema and their parents. More specifically, we predict:

* There will be a reduction in negative parental idiosyncratic measures of stress throughout the intervention phase, in comparison to baseline phase, that will be maintained in the follow-up phase.
* There will be an improvement in positive parental idiosyncratic measures of stress during the intervention phase in comparison to baseline phase that will be maintained in the follow-up phase.
* There will be a significant increase in levels of mindful parenting following the intervention phase, in comparison to baseline phase, that will be maintained in the follow-up phase.
* There will be a significant decrease in levels of parental stress at end of intervention phase compared to baseline phase that will be maintained in the follow-up phase.
* There will be a significant increase in parental quality of life and paediatric quality of life at the end of intervention phase compared to baseline phase that will be maintained in the follow-up phase .
* There will be a significant improvement in psoriasis severity and itch at the follow-up phase compared to the baseline phase.

ELIGIBILITY:
Child inclusion criteria:

* Received a diagnosis of psoriasis or eczema from a medical professional
* Aged 4-16 years
* Fluent English speaker
* Psoriasis or eczema is the primary health concern

Parent inclusion criteria:

* Parent of child (aged four to 16 years old) with psoriasis or eczema
* Aged 16 or over
* Self-identifies as experiencing stress due to the child's skin condition
* Fluent English Speaker
* Able and willing to attend 9 group sessions
* Willing to commit sufficient time to carrying out the practice (e.g. at home)
* Willing to respond to daily brief text messages

Child exclusion criteria:

- N/A

Parent exclusion criteria:

* Active thoughts of suicide
* Active thoughts of self-harm
* Engaging in, or about to start, psychological therapy during the study period
* Previously attended a mindful parenting group
* Recent severe life events such as deliberate self-harm, hospital admission, or psychotic episode (last 12 months)
* Experiencing physical pain or problems that may be worsened by yoga exercises.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Change in parenting stress (idiosyncratic measure) | Daily for 20 weeks (baseline-intervention-follow-up)
  The primary outcome measures for the proposed study are idiosyncratic measures of stress which will be assessed daily by text message. Participants will be asked to identify one stress-related positive target (something the participant would like to improve) and one negative target (something the participant would like to reduce). Participants will respond to the daily text messages with a score on a 0-100 scale.

SECONDARY OUTCOMES:
Demographic information | 1-time point (baseline period)
  Parents will be asked to provide information about their age, gender, ethnicity, relationship to child, employment status, marital status, education level, child's age, and child's gender.
Mindful parenting | 4 time-points. Baseline (beginning of study), beginning of intervention (2 weeks later) end of intervention (8 weeks later) follow-up (8 weeks later)
  The Interpersonal Mindfulness in Parenting scale (IM-P; Duncan, 2007) will be used to ascertain the level of mindful parenting of the parents. This self-report questionnaire measures affective, cognitive and attitudinal aspects of parent-child relationships. There are 10 items covering one higher order mindful parenting factor and four first-order factors: 1) present-centered attention in parenting; 2) present-centered emotional awareness in parenting; 3) non-reactivity/low-reactivity in parenting; and 4) non-judgmental acceptance in parenting. Items are rated on five-point Likert scales (from "never true" to "always true").
Parental Stress | 4 time-points. Baseline (beginning of study) beginning of intervention (2 weeks later), end of intervention (8 weeks later), follow-up (8 weeks later)
  The Parenting Stress Index - Short Form (PSI-SF; Abidin, 1995) will be used to assess parental stress. This 36-item self-report measure assesses parental stress over three factors (parental distress, dysfunctional parent-child interactions, and difficult child) and one total stress factor (Abidin, 2012). Items are rated on a 5-point Likert scale (from "strongly agree" to "strongly disagree")
Parental Anxiety | 4 time-points. Baseline (beginning of study), beginning of intervention (2 weeks later), end of intervention (8 weeks later), follow-up (8 weeks later)
  The Generalised Anxiety Disorder Questionnaire (GAD-7; Spitzer, Kroenke & Williams, 2006) is a 7-item self-report scale to measure generalized anxiety symptoms. Items are rated on a 4-point Likert scale (from "not at all" to "nearly everyday").
Parental Depression | 4 time-points. Baseline (beginning of study), beginning of intervention (2 weeks later), end of intervention (8 weeks later), follow-up (8 weeks later)
  The Patient Health Questionnaire (PHQ-9; Spitzer, Kroenke, & Willams, 1999) is a 9-item questionnaire assessing symptoms of depression. Items are rated on a 4-point Likert scale (from "not at all" to "nearly everyday")
General Stress | 5 time-points. Screening interview (pre-study), baseline (beginning of study, approx. 2-4 weeks later), beginning of intervention (2 weeks later), end of intervention (8 weeks later), follow-up (8 weeks later)
  The stress subscale of the Depression Anxiety and Stress Scale (DASS-21: Lovibond & Lovibond, 1995) will be used to assess general stress levels of parents. Items are rated on 4-point Likert scale (from "never" to "almost always").
Parental quality of life | Baseline (beginning of study), beginning of intervention (2 weeks later), end of intervention (8 weeks later), follow-up (8 weeks later)
  The Family Dermatology Life Quality Index (FDLQI: Basra, Su-Ho, & Finlay, 2007) will be used to measure parental quality of life. This self-report measure comprises 10 items assessing a range of ways that a family member's skin condition may impact upon an individual's quality of life, covering two factors (psychosocial impact and physical impact). Items are rated on a 4-point Likert scale (ranging from "not at all" to "very much").
Paediatric quality of life | Baseline (beginning of study), beginning of intervention (2 weeks later), end of intervention (8 weeks later), follow-up (8 weeks later)
  The Children's Dermatology Life Quality Index (CDLQI: Lewis-Jones & Finlay, 1995) will be used to assess paediatric quality of life. This self-report measure is completed by the child, and comprises 10-items assessing a range of ways that a child's skin condition may impact upon their quality of life, covering 6 areas (symptoms and feelings, leisure, school or holidays, personal relationships, sleep, treatment). Items are rated on a 4-point Likert scale (ranging from "not at all" to "very much").
Paediatric psoriasis/eczema severity | 2 time-points. Baseline (beginning of study), follow-up (18 weeks later)
  Children will be asked to indicate the itch intensity of the psoriasis/eczema, on a 10-point scale (from "not at all itchy" to "the worst itchy imaginable")
Paediatric psoriasis/eczema itch intensity | 2 time-points. Baseline (beginning of study), follow-up (18 weeks later)
  Children will be asked to indicate the itch intensity of the psoriasis/eczema, on a 10-point scale (from "not at all bad/severe" to "extremely bad/severe").

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire
  - The University of Sheffield, Sheffield, South Yorkshire
  - Sheffield Children's Hospital, Sheffield, South Yorkshire
  - Doncaster Royal Infirmary, Doncaster
  - Rotherham Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abidin, R. R. (1995). Parenting stress index 3rd edition: Professional manual. Psychological Assessment Resources, Inc, Odessa, TX.
- [Background] Abidin R. R. (2012) Parenting Stress Index. Odessa, FL: Psychological Assessment Resources.
- [Background] Basra MK, Sue-Ho R, Finlay AY. The Family Dermatology Life Quality Index: measuring the secondary impact of skin disease. Br J Dermatol. 2007 Mar;156(3):528-38. doi: 10.1111/j.1365-2133.2006.07617.x. PMID 17300244
- [Background] Bögels, S., & Restifo, K. (2013). Mindful parenting: A guide for mental health practitioners. Springer Science & Business Media.
- [Background] Duncan, L. G. (2007). Assessment of mindful parenting among parents of early adolescents: Development and validation of the Interpersonal Mindfulness in Parenting scale. The Pennsylvania State University.
- [Background] Kabat-Zinn, J. (1990). Full catastrophe living. New York: Bantam Doubleday Dell.
- [Background] Lewis-Jones MS, Finlay AY. The Children's Dermatology Life Quality Index (CDLQI): initial validation and practical use. Br J Dermatol. 1995 Jun;132(6):942-9. doi: 10.1111/j.1365-2133.1995.tb16953.x. PMID 7662573
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171